CLINICAL TRIAL: NCT05788315
Title: The Influence of the Cultural Formulation Interview on Cultural Empathy and the Therapeutic Work Alliance in Clients With a Migration Background and Their Informants
Brief Title: The Influence of the Cultural Formulation Interview on Therapeutic Work Alliance
Acronym: CFITWA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tilburg University (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Alma Brand, Principal Investigator, Tilburg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 6390039231
Record Dates: First submitted 2023-03-01; First posted 2023-03-28 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Therapeutic Alliance; Empathy
Keywords: Cultural Formulation Interview; Therapeutic Working Alliance; Cultural Empathy; Migrants; Migratory Background; Ethnicity

STUDY DESIGN:
Intervention Model Description: This study will be set up as a cluster RCT among CMBs who are admitted to outpatient care at the four participating mental healthcare centers.
Who Masked: Participant
Masking Description: One half of the participants will be assessed using the Cultural Formulation Interview The other half will be assessed using the standard practice intake
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cultural Formulation Interview (Experimental): The 16 semi-structured questions of the CFI cover the cultural definition of the problem, cultural perception of its cause, context and support, cultural aspects of coping, and past and present help-seeking behavior. The CFI informant version consists of 17 questions about the same themes. The CFI aims to bridge cultural differences by explicitly asking about the client's cultural background and its influence on the presented problems
  Interventions: Other: Cultural Formulation Interview
- Standard Care (Active Comparator): Standard intake and care
  Interventions: Other: Cultural Formulation Interview

INTERVENTIONS:
Other: Cultural Formulation Interview — The Cultural Formulation Interview will be used at the start of treatment in the intervention group against a standard practice intake in the control group.

SUMMARY:
The increased cultural diversity in client populations in mental healthcare settings led to the addition of the Cultural Formulation Interview (CFI) in the Diagnostic and Statistical Manual for Mental Disorders (DSM-5). The CFI aims to clarify clients' vision, experiences, and context to improve communication about cultural backgrounds, increase mutual understanding and rapport, and prevent cultural misunderstandings. Empirical evidence of this effect in clinical practice is still lacking.

This study investigates whether the CFI influences the therapeutic working alliance between a client with a migration background and a clinician, and the informant version of the CFI (CFI-I) influences the relationship between a client's informant and a clinician, focusing on the role of perceived cultural empathy as moderator, or mediator in this interaction.

A Cluster-Randomized Controlled Trial (RCT) will be performed among clients with a migratory background in four mental healthcare centers in the Netherlands. The participants in this study are adults with a migratory background, aged 18 years and older, their informants, and clinicians.

Participants were randomly assigned into two groups. In the intervention group, the CFI and CFI-Informant version (CFI-I) were used shortly after admission and intake, and the control group received a clinical assessment as usual. Included informants were assessed with the CFI-I or hetero-anamneses by the participating clinicians.

The main outcome measure is the work alliance between clients and their clinicians. This will be evaluated using the Work Alliance Questionnaire. Perceived cultural empathy as a potential mediator or moderator will be measured with the Barrett-Lennart Relationship Inventory among clients and informants, and the Scale of Ethnocultural Empathy among clinicians.

The clients and informants will be randomly assigned to the intervention group or the control group. They will all fill out a questionnaire about perceived cultural empathy after the first, and two questionnaires about work alliance, and perceived cultural empathy after five treatment sessions. The clinicians will perform the clinical assessments with or without the CFI and fill out a questionnaire about self-perceived cultural empathy after the first session and two questionnaires about work alliance and cultural empathy after a maximum of five given treatments. There is no physical, behavioral, or medical intervention included in the research protocol.

DETAILED DESCRIPTION:
Mental health care for clients with a migratory background (CMB) is less effective than for clients without a migration background. For instance, CMB show higher rates of dropout, have longer care trajectories, show lower treatment effects, and are more frequently forced into clinical care. Part of the explanation for this might be higher thresholds to seek help and treatment mismatches due to a lack of adaptation of the diagnostic and treatment methods to the client's needs. Despite the positive fact that CMB have more frequently sought help over the past years, the drop-out remains high because CMB care needs are often not met. To make amends for this problem, the need for clinical instruments emerged to clarify the influence of cultural aspects in diagnostics. This led to the first draft of the Cultural Formulation Interview (CFI), which was added to the DSM-5, aiming for clinicians to gain more insight into the illness perspectives of CMB when using the instrument. This semi-structured interview contains 16-17 questions that aim to bridge gaps between differences in cultural referential frameworks of CMB and clinicians which may improve healthcare for CMB. The CFI enhances communication about culture, which increases mutual understanding and rapport based on interest and better apprehension of the client's cultural background aiming to prevent cultural misunderstandings. Research shows that the use of the CFI positively influences communication between CMB and clinicians. Empathy is crucial in this communication because an empathic clinician will better understand the client's problems and come up with more adequate diagnoses, which benefit the CMB.

Empathy refers to the emotional and cognitive reactions to the observed experiences of someone else. Empathy is defined as the accurate acknowledgment of the internal reference framework of another person integrated with the emotional components and implication to be the other, by putting oneself into someone else's position. Empathy is an important ingredient for building relationships between clients and clinicians. This is even more important when practicing effective culture-sensitive psychotherapy. Cultural empathy is the capacity to identify with the feelings, thoughts, and behavior of people with a different cultural background than one's own by listening and hearing beyond spoken words and bridging cultural differences. The level of cultural empathy can influence the strength and quality of a therapeutic relationship, which is also known as work alliance. The strength of a working alliance depends on the level of agreement with the treatment goals and given tasks within the therapy, and the affective quality of the relationship between the CMB and the clinician.

In an exploratory qualitative study during the implementation phase of the CFI-test version, tentative optimistic signs regarding satisfaction and clarity were found, whilst an earlier study reported resistance against the implementation of the CFI from both CMB and clinicians' perspectives. No research has been done to examine CFI use concerning work alliance and cultural empathy. The need to perform a random controlled trial (RCT) emerged because part of the CFI questions was experienced as problematic. Despite previous findings, it is expected that using the CFI with CMB strengthens the working alliance between CMB and clinicians, either mediated or moderated by cultural empathy. Outcomes could help to improve mental healthcare by stronger work alliance and lower drop-out rates through better communication, understanding, and empathy between CMB and clinicians.

This study empirically investigates whether using the CFI increases the clients' and informant's sense of being understood within their cultural context, and thus encounter cultural empathy and whether due to perceived cultural empathy they experience a stronger working alliance with their clinician. Outcomes might convince clinicians of the usefulness and relevance of the structural use of the CFI in clinical practice, especially when this proves to increase perceived (cultural) empathy and strengthen work alliance. It is expected that a culture-sensitive working alliance between CMBs, informants, and clinicians could be a crucial aspect in reducing the high drop-out and relatively low effect on mental health care for first and second-generation migrants. The central research question in this study is: To what extent do the use of the CFI for CMB and their informants change their work alliance with clinicians? This change could be moderated (changed in strength and direction) or mediated (explained) by cultural empathy. It is hypothesized that the use of the CFI will improve the therapeutic working alliance moderated (strengthened) by cultural empathy.

ELIGIBILITY:
Inclusion Criteria:

* Participants can be included if they:

  * Are older than 18 years.
  * Have a first or second-generation migration background.
  * Are newly and voluntarily admitted to outpatient mental health care (to avoid bias by forced admissions, which might jeopardize work alliances because of the complex nature of the presented mental health problems).
  * Are capable to communicate their perspective, context, and expectations regarding the provided care.

Exclusion Criteria:

* Participants will be excluded when:

  * They are mentally incapable of administering questionnaires or reflecting on their personal situation.
  * They are incapable to communicate their perspective, context, and expectations regarding the care provided in this research project.
  * They suffer acute mental illnesses.
  * They abuse substances (for example: alcohol and/or drugs).

    * The absence of or objection against including an informant is no exclusion criterion.
    * There are no in- or exclusion criteria around diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Therapeutic Work Alliance (participants) | 3 months
  The Work Alliance Inventory (WAI-12) will be used to measure work alliance among participants. The WAI-12 measures the strength of the working alliance with 12 items utilizing a 5-point Likert scale. The minimum score is 0, the maximum score is 48. Higher scores indicate a stronger working alliance.
Therapeutic Work Alliance (clinicians) | 3 months
  The Work Alliance Inventory (WAI-therapist version) will be used to measure work alliance among clinicians. The WAI for therapists measures the strength of the working alliance with 36 items utilizing a 5-point Likert scale. The minimum score is 0, the maximum score is 180. Higher scores indicate a stronger working alliance.

SECONDARY OUTCOMES:
Cultural Empathy (participants) | 1 week and 3 months
  The Barret-Lennard Relationship Index (BLRI) is used to measure perceived empathy in CMB and informants. The 64-item self-to-other version consists of items such as: '[clinician's name] cares for me', '[clinician's name] just tolerates me', and '[clinician's name] is truly interested in me'. The items are scored on a 6-point Likert scale (-3, -2, -1, 1, 2, 3). The minimum score is -192, and the maximum score is 192. Higher scores indicate a higher level of perceived cultural empathy. This scale will be administered twice.
Cultural Empathy (clinicians) | 1 week and 3 months
  The Scale of Ethnocultural Empathy (SEE) is used to measure the clinician's level of cultural empathy. The 31 items are scored in an online survey on a 6-point Likert scale. The minimum score is 0 and the maximum score is 155. Higher scores indicate a higher level of cultural empathy. This scale will be administered twice.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Braakman, Prof., Study Director — Tilburg University
Locations (1):
- Onderzoek Consortium Samen Sterker, Tilburg, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
A DMP has been written, checked, and uploaded on DMP Online
Supporting Information: SAP, CSR, Analytic Code
Time Frame: Immediately after the end of the study during 10 years
Access Criteria: Data will be anonymous and stored in TiU Dataverse using DDI. We are contemplating using an archive or repository.
URL: https://dmponline.dcc.ac.uk/plans/110742